CLINICAL TRIAL: NCT04977830
Title: New Strategies for Pulmonary Assessment in Spinal and Chest Wall Deformity
Brief Title: Pulmonary Assessment in Thoracic Insufficiency Syndrome Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Cahill, MD (Other)
Collaborators: Xemed LLC (Industry)
Responsible Party: Sponsor-Investigator, Patrick Cahill, MD, Attending physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-017344
Record Dates: First submitted 2021-07-14; First posted 2021-07-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Insufficiency Syndrome
Keywords: Hyperpolarized MRI; Dynamic Lung MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Thoracic Insufficiency Group (Other): Thoracic insufficiency syndrome patients undergoing surgery
  Interventions: Device: Xenon-129

INTERVENTIONS:
Device: Xenon-129 — Patients will undergo a hyperpolarized MRI with administered Xenon gas

SUMMARY:
Thoracic insufficiency syndrome (TIS) is a complex condition that involves chest wall deformities that can affect normal breathing and lung growth. In most cases, children with TIS are also born with spine disorders such as scoliosis. The inability of the thorax to support normal respiration or lung growth can cause respiratory distress and even mortality. Investigators aim to validate MRI imaging sequences to use as an assessment tool for pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 6 to 18 years old diagnosed with thoracic insufficiency syndrome who are undergoing surgery

Exclusion Criteria:

* patients not diagnosed with thoracic insufficiency syndrome

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Analyze volume of lungs at end-inspiration and end-expiration | up to 2 years
  Investigators will analyze lung volume at end-inspiration and end-expiration will be assessed by performing a thoracic dynamic magnetic resonance imaging scan; measured in total volume units (mL)
Xenon-129 MRI Ventilation Maps | up to 2 years
  Xenon-129 MRI will be completed to reveal unventilated regions of the lungs where the gas cannot reach after being inhaled due to restrictions of the airways.

SECONDARY OUTCOMES:
oxygen partial pressure (PAO2) maps | up to 2 years
  Oxygen partial pressure (PAO2) maps will be extracted from 129Xe MRI maps in a single breath-hold. Regions of the lungs that show abnormal PAO2 values are susceptible of improper ventilation or gas exchange.
Forced vital capacity (FVC) | up to 2 years
  Forced vital capacity will be extracted from the computer-automated dynamic lung MRI software.
Forced expiratory volume (FEV1) | up to 2 years
  Forced expiratory volume data will be extracted from the computer-automated dynamic lung MRI software to assess the volume of air forced from the lungs
Xenon-129 MRI apparent diffusion coefficient (ADC) maps | up to 2 years
  Apparent diffusion coefficient (ADC) maps are extracted from the Xenon-129 MRI from a single breath-hold pulse sequence.
total lung capacity | up to 2 years
  Total lung capacity will be extracted from the computer-automated dynamic lung MRI software.
functional residual capacity (FRC) | up to 2 years
  functional residual capacity data will be extracted from the computer-automated dynamic lung MRI software to measure the volume in the lungs at the end of passive expiration

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cahill, MD, Principal Investigator — Children's Hopsital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States